CLINICAL TRIAL: NCT01871857
Title: 7% Hypertonic Saline for Acute Bronchiolitis: A Randomized Controlled Trial
Brief Title: 7% Hypertonic Saline for Acute Bronchiolitis
Acronym: HS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Le Bonheur Children's Hospital (Other)
Responsible Party: Principal Investigator, Jonathan Jacobs, Pediatric Emergency Physician, Le Bonheur Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LCH
Record Dates: First submitted 2013-05-29; First posted 2013-06-07 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Acute Bronchiolitis
MeSH Terms: interventions — Saline Solution, Hypertonic; Epinephrine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal saline and epinephrine (Active Comparator): 0.9 % saline with 0.5 ml of 1:1000 epinephrine inhalation
  Interventions: Drug: Normal saline and epinephrine
- Hypertonic saline and epinephrine (Experimental): 3 ml 7% saline with 0.5 ml of 1:1000 epinephrine inhalation
  Interventions: Drug: Hypertonic saline and epinephrine

INTERVENTIONS:
Drug: Hypertonic saline and epinephrine
  Arms: Hypertonic saline and epinephrine
Drug: Normal saline and epinephrine
  Arms: Normal saline and epinephrine

SUMMARY:
Research suggests that hypertonic saline may improve mucous flow in infants with acute bronchiolitis. Data suggest a trend favoring reduced length of hospital stay and improved pulmonary scores with increasing concentration of nebulized solution to 3% and 5% saline as compared to 0.9% saline mixed with epinephrine. To our knowledge, 7% hypertonic saline has not been previously investigated. OUr hypothesis was that 7% hypertonic saline would improve bronchiolitis severity scores and admission rate.

DETAILED DESCRIPTION:
Study design A double-blinded, randomized, comparative, controlled trial was conducted in the ED of an urban tertiary care center, with an annual census of 70,000 patient visits. The Institutional Review Board approved the study.

Patient selection Informed consent was obtained from a parent or legal guardian of each patient enrolled in the study. Patients age 6 weeks to ≤ 18 months presenting to the ED between October and March over a 2-year period (2010-2012) with bronchiolitis (defined as viral respiratory illness and first episode of wheeze) and a BSS score of ≥ 4 were eligible for the study. Exclusion criteria were a previous history of wheezing; diagnosis of asthma; any use of bronchodilators within 2 h of presentation; gestational age ≤ 34 weeks; history of congenital heart disease, chronic pulmonary or chronic renal disease; oxygen saturation of ≤ 85% at the time of recruitment; severe disease requiring intensive care unit admission, or inability to obtain informed consent. Depending on the availability of the principal investigator (a pediatric emergency medicine fellow), a convenience sample was used to recruit patients. The ED physicians and staff were notified of the fellow's hours of availability by way of a call schedule that was posted in the ED.

Study protocol Eligible patients were randomized to one of two groups in blocks of 10. The control group received an aerosol of 0.5 ml of 2.25% racemic epinephrine with 3 ml of 0.9% saline, and the study group received 0.5 ml of 2.25% racemic epinephrine with 3 ml of 7% HS.

The treating clinician in the ED contacted the principal investigator within an hour of an eligible patient's arrival. The pharmacy department maintained a box in the ED holding sequentially numbered, previously randomized concealed envelopes containing either the study (7% HS) or control (0.9% saline) medication. After initial screening and assessment and after consent was obtained, the patient was administered the medication via nebulization driven by 6 L/min O2 flow. Research personnel, the treating physician, and staff who performed the BSS were kept blinded throughout the process. Bronchiolitis severity scores were recorded prior to administering aerosols, after administering the aerosol, and again once the treating clinician determined the final disposition of the patient.

After a 4-h observation period, the treating clinician determined patient disposition. If admitted, the patient continued to receive aerosols containing the same designated medication every 6 h until discharge or 24 h after the admission. Bronchiolitis severity scores were obtained before and after each treatment. A standardized data sheet was completed after enrollment and during each patient's stay in the ED or inpatient ward. Any co-interventions such as additional bronchodilators, supplemental oxygen, intravenous fluids, or deep nasal suction were at the discretion of the treating clinician. The clinician was free to withdraw the patient from the study if clinical deterioration warranted escalation of care or if adverse effects related to the medication were observed.

Outcome measures The BSS is an objective respiratory assessment tool that has been previously validated (Table 1).14 We used a modified BSS, which is used in our institution since 2006, to assess severity of illness in acute bronchiolitis. (Table 2) A change in the modified BSS was the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 6 weeks to ≤ 18 months
* Diagnosed with bronchiolitis (defined as viral respiratory illness and first episode of wheeze)
* BSS score of ≥ 4

Exclusion Criteria:

* A previous history of wheezing;
* diagnosis of asthma;
* any use of bronchodilators within 2 h of presentation
* gestational age ≤ 34 weeks
* history of congenital heart disease
* chronic pulmonary or chronic renal disease
* oxygen saturation of ≤ 85% at the time of recruitment
* severe disease requiring intensive care unit admission
* inability to obtain informed consent

Ages: 6 Weeks to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2010-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in Bronchiolitis Severity Score | Baseline and up to 24 hours of hospital stay
  Bronchiolitis severity scores were recorded prior to administering aerosols, after administering the aerosol, and again once the treating clinician determined the final disposition of the patient.
  After a 4-h observation period, the treating clinician determined patient disposition. If admitted, the patient continued to receive aerosols containing the same designated medication every 6 h until discharge or 24 h after the admission. Bronchiolitis severity scores were obtained before and after each treatment.

SECONDARY OUTCOMES:
Admission rate | For approximately 2 yrs, the duration of the study
  Secondary outcome measures included hospitalization rate, discharge rate at 23 h (observation status), and length of hospital stay. These are a composite of measures reflecting impact of hypertonic saline on in-patient metrics

CONTACTS AND LOCATIONS:
Overall Officials: Jay Pershad, MD, Study Director — Le Bonheur Children's Hospital
Locations (1):
- Le Bonheur Children's Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Jacobs JD, Foster M, Wan J, Pershad J. 7% Hypertonic saline in acute bronchiolitis: a randomized controlled trial. Pediatrics. 2014 Jan;133(1):e8-13. doi: 10.1542/peds.2013-1646. Epub 2013 Dec 16. PMID 24344111